CLINICAL TRIAL: NCT05184907
Title: Effects of Remote Motivational Enhancement on Engagement in Buprenorphine Treatment
Brief Title: Effects of RME on Engagement in Buprenorphine Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge Health Alliance (Other)
Collaborators: University of South Florida (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHA-IRB-21-22-29; R01CE003039 (NIH)
Record Dates: First submitted 2021-11-24; First posted 2022-01-11 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Opioid Use Disorder; Behavioral Symptoms; Psychiatric or Mood Diseases or Conditions
MeSH Terms: conditions — Opioid-Related Disorders; Behavioral Symptoms

STUDY DESIGN:
Intervention Model Description: RME (1-3 sessions) versus information alone
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RME Intervention Arm (Experimental): Participants will discuss the results of their CAT-MH, BAM, and PSS with a coach trained in motivational interviewing with 14 days of study randomization. Based on these results, the coach will help to identify behavior change goals, resolve ambivalence, amplify activation, explore their options, and empower the participant toward taking action to obtain appropriate support services tailored to their individual issues and concerns. The number of RME sessions will range from 1-3, determined by the participant's level of activation and desire to engage in additional sessions, as well as the number of challenges identified in their initial session or determined by their CAT-MH results. Participants will be sent a link at the end of week 1 with the aim to complete an action plan questionnaire, in which they will be asked to describe up to 3 action plan goals (in mental health, social services, and stress reduction/mental wellness categories).
  Interventions: Behavioral: Remote Motivational Enhancement (RME) Intervention Arm
- Information Only Arm (Active Comparator): Participants randomized to the information-only arm will have their CAT-MH, BAM, and PSS screening report results sent to their primary B/N prescriber and will encouraged to set up an appointment with their prescriber within 14 days to discuss the results. Participants will be sent a link at the end of week 1 with the aim to complete an action plan questionnaire, in which they will be asked to describe up to 3 action plan goals (in mental health, social services, and stress reduction/mental wellness categories).
  Interventions: Other: Information Only

INTERVENTIONS:
Behavioral: Remote Motivational Enhancement (RME) Intervention Arm — Participants will discuss the results of their CAT-MH, BAM, and PSS with a coach trained in motivational interviewing within 14 days of study randomization. Based on these results, the coach will help to identify behavior change goals, resolve ambivalence, amplify activation, explore their options, and empower the participant toward taking action to obtain appropriate support services tailored to their individual issues and concerns. The number of RME sessions will range from 1-3, determined by the participant's level of activation and desire to engage in additional sessions, as well as the number of challenges identified in their initial session or determined by their CAT-MH results. Participants will be sent a link at the end of week 1 with the aim to complete an action plan questionnaire, in which they will be asked to describe up to 3 action plan goals (in mental health, social services, and stress reduction/mental wellness categories).
  Arms: RME Intervention Arm
Other: Information Only — Participants randomized to the information-only arm will have their CAT-MH, BAM, and PSS screening report results sent to their primary B/N prescriber and will encouraged to set up an appointment with their prescriber within 14 days to discuss the results. Participants will be sent a link at the end of week 1 with the aim to complete an action plan questionnaire, in which they will be asked to describe up to 3 action plan goals (in mental health, social services, and stress reduction/mental wellness categories).
  Arms: Information Only Arm

SUMMARY:
The investigators will conduct a Randomized Controlled Trial (RCT) comparing the Remote Motivational Enhancement (RME) coaching sessions + MindWell screenings arm to an Information-only + MindWell screenings arm on early engagement in treatment support services, as measured by overall action plan initiation.

DETAILED DESCRIPTION:
In an effort to assess and address patients' mental health needs, Cambridge Health Alliance has developed an innovative screening program (MindWell) using electronic computerized adaptive testing that will be used among telemedicine patients with opioid use disorder prescribed buprenorphine by Bicycle Health to evaluate needs related to mental health (CAT-MH) and social determinants of health (CAT-SDOH), as well as for stress (Perceived Stress Scale-PSS) and addiction (Brief Addiction Monitor- BAM). This automated screening with adaptive testing helps to identify those who need social services support (e.g. housing, legal, immigration, financial, food, transportation, etc.) or need further comprehensive mental health evaluation and treatment.

Remote Motivational Enhancement (RME) sessions provide telehealth coaching sessions based on motivational interviewing (MI), which is a collaborative, goal-oriented style of communication designed to resolve ambivalence and strengthen intrinsic motivation for a person's commitment to behavior change by eliciting their own reasons for change in an environment of acceptance and compassion. It is an evidence-based and standardized approach that has demonstrated consistently positive clinical outcomes for engagement in wellness, healthcare, and addiction treatment, including effectively improving medical regimen adherence.

This study will randomize Bicycle Health patients prescribed Buprenorphine/Naloxone (B/N) who have been screened the MindWell system to receive either standard care reviewing their screening results with their prescriber or they will receive the opportunity to additionally receive up to 3 RME sessions within a 14 day period. This study investigates the effects of the RME intervention on early engagement in psychosocial aspects of B/N telehealth treatment, rates of opioid overdose, and B/N treatment retention. This study will assess the impact of RME sessions on participants' capacity to achieve behavior change goals related to their individual SDOH needs, mental health symptoms, and/or wellness in OUD recovery goals.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Meets DSM-IV criteria for opioid dependence or DSM-V criteria for opioid use disorder
* Current patient enrolled in Bicycle Health's buprenorphine treatment program
* Ability to provide informed consent
* Access to the internet and an electronic device to attend remote coaching sessions via videoconferencing and complete online assessments
* Sufficient English fluency to understand study procedures and assessments
* Completion of the CAT-MH screening modules, BAM, and PSS measures (through CHAMindWell and Bicycle Health's service implementation project)

Exclusion Criteria:

* Non-English speaking
* Reporting active homicidal or suicidal ideation
* Exhibits signs of active mania or psychosis
* Expected incarceration in next 12 weeks (those that are incarcerated during the study will be withdrawn from the study)
* Prisoners
* Unable or unwilling to use a mobile device
* Has a medical contraindication to BUP
* Unable to complete screening and baseline assessments
* Unstable medical illness that could lead to an expected hospitalization in the next 12 weeks
* Third-trimester pregnancy (if a pregnant participant plans to deliver within 12 weeks of study consent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-08-02 (Actual)

PRIMARY OUTCOMES:
Engagement through Action Plan Initiation | 4 weeks
  1. To examine the effects of RME sessions versus information alone on early engagement in treatment support services as measured by the Action Plan Initiation Survey (APIS-5) with a score of 5-7 representing action plan initiation.

SECONDARY OUTCOMES:
Number of Self-Reported and Clinic-Reported Opioid Overdose | 12 weeks
  To examine the effect of RME versus information alone on the number of self-reported (with and without naloxone administered) and clinic-reported opioid overdoses throughout the 12 weeks of the study.
B/N Treatment Retention | 24 weeks
  To examine the effect of RME versus information alone on retention in buprenorphine OUD treatment with an active prescription at 24 weeks as assessed by an active prescription with Bicycle Health in the past 30 days.
Brief Addiction Monitor Scale | 12 weeks
  To examine the effect of RME versus information alone on change in Brief Addiction Monitor (BAM) subscale scores from 0 to 12 weeks.
  1. Drug Use (lower is better outcome)
  2. Risk Factors (lower is better outcome) (>12 is considered high risk)
  3. Protective Factors (higher is better outcome) (<12 is considered high risk)

OTHER OUTCOMES:
Action Plan Initiation: Social Service Engagement | 12 weeks
  To examine the effects of RME sessions vs. information alone on early engagement in types of treatment support services as measured by initiation in the social service subtype of treatment engagement.
  Initiation and engagement of support services for issues related to social determinants of health as measured by action plan initiation self-report at 4 weeks and/or reported appointment with social service professionals within 12 weeks.
Action Plan Initiation: Mental Health Engagement | 12 weeks
  To examine the effects of RME sessions vs. information alone on early engagement in types of treatment support services as measured by initiation in the mental health subtype of treatment engagement.
  Self-reported initiation and engagement with mental health services for psychiatric symptoms as measured by action plan initiation self-report at 4 weeks and reported appointment with mental health professionals within 12 weeks.
Action Plan Initiation: Wellness/Stress Reduction Engagement | 12 weeks
  To examine the effects of RME sessions vs. information alone on early engagement in types of treatment support services as measured by initiation in the wellness/stress reduction subtype of treatment engagement.
  Self-reported initiation of mental wellness/stress reduction services by action plan initiation self-report at 4 weeks and reported appointment with mental health professionals within 12 weeks.
Changes in Substance Use Risk | 12 weeks
  To examine a change in CAT-MH-SUD risk scores from 0 to 12 weeks. CAT-MH-SUD is computerized adaptive testing with a normalized score ranging from 0-100 (lower scores are better outcome).
Changes in Social Vulnerability | 12 weeks
  To examine a change in CAT-MH-SDOH scores from 0 to 12 weeks. CAT-MH-SDOH is computerized adaptive testing with a normalized score ranging from 0-100 (higher scores are better outcome).
Changes in Anxiety | 12 weeks
  To examine a change in CAT-MH-Anxiety scores from 0 to 12 weeks. CAT-MH-Anxiety is computerized adaptive testing with a normalized score ranging from 0-100 (lower scores are better outcome).
Changes in Depression | 12 weeks
  To examine a change in CAT-MH-Depression scores from 0 to 12 weeks. CAT-MH-Depression is computerized adaptive testing with a normalized score ranging from 0-100 (lower scores are better outcome).
Changes in Psychosis | 12 weeks
  To examine a change in CAT-MH-Psychosis scores from 0 to 12 weeks. CAT-MH-Psychosis is computerized adaptive testing with a normalized score ranging from 0-100 (lower scores are better outcome).
Changes in PTSD symptoms | 12 weeks
  To examine a change in CAT-MH-PTSD scores from 0 to 12 weeks. CAT-MH-PTSD is computerized adaptive testing with a normalized score ranging from 0-100 (lower scores are better outcome).
Changes in Mania/Hypomania | 12 weeks
  To examine a change in CAT-MH-Mania/Hypomania scores from 0 to 12 weeks. CAT-MH-M/HM is computerized adaptive testing with a normalized score ranging from 0-100 (lower scores are better outcome).
Changes in ADHD symptoms | 12 weeks
  To examine a change in CAT-MH-ADHD scores from 0 to 12 weeks. CAT-MH-ADHD is computerized adaptive testing with a normalized score ranging from 0-100 (lower scores are better outcome).
Changes in Level of Intrinsic Motivation | 4 and 12 weeks
  To examine between-group differences in APA-10 scores at weeks 4 and 12 (Higher levels represent increased intrinsic motivation). (Assessing self-efficacy and self-actualization as indicators of intrinsic motivation in accordance with the self-determination theory.)
Changes in Treatment Services Needed and Received | 12 weeks
  To examine between-group differences in the change in Treatment Services Needed and Received scores from baseline to week 12 (Each item represents a service that participants indicate needing and/or receiving over the past two weeks. The measure includes separate scales for assessing the need and receipt of medical services (6 items), alcohol / drug services (16 items), psychological / emotional services (18 items), psychiatric crisis services (8 items), and other services (22 items). The amount of unmet service needs is calculated by subtracting the number of services received in each area from the number needed in that respective area.)

CONTACTS AND LOCATIONS:
Overall Officials: Zev Schuman-Olivier, MD, Principal Investigator — Cambridge Health Alliance; Kathleen Moore, PhD, Principal Investigator — University of South Florida
Locations (1):
- Cambridge Health Alliance, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data related to our outcome measures will be included in the IPD sharing plan, in addition to our study protocol, informed consent, and analytic plan.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication and within 12 months of completion of the analysis of study primary aims, anonymous and de-identified data will be made available at the Open Science Framework (http://osf.io/) and/or Harvard Dataverse (https://dataverse.harvard.edu/) so that other investigators can verify or follow-up on the reported analyses.
Access Criteria: Anonymous and de-identified data will be stored on the Open Science Framework website (http://osf.io/) and/or Harvard Dataverse to be made available to other researchers to verify the research results. Before publication, only USF and CHA investigators will have direct access to the data, and only the CHA HERLab or CHA Center for Mindfulness and Compassion investigators will have access to the analyses.

REFERENCES:
- [Background] Achtyes ED, Halstead S, Smart L, Moore T, Frank E, Kupfer DJ, Gibbons R. Validation of Computerized Adaptive Testing in an Outpatient Nonacademic Setting: The VOCATIONS Trial. Psychiatr Serv. 2015 Oct;66(10):1091-6. doi: 10.1176/appi.ps.201400390. Epub 2015 Jun 1. PMID 26030317
- [Background] Drake C, Yu J, Lurie N, Kraemer K, Polsky D, Chaiyachati KH. Policies to Improve Substance Use Disorder Treatment With Telehealth During the COVID-19 Pandemic and Beyond. J Addict Med. 2020 Sep/Oct;14(5):e139-e141. doi: 10.1097/ADM.0000000000000727. PMID 32826619
- [Background] Gibbons RD, deGruy FV. Without Wasting a Word: Extreme Improvements in Efficiency and Accuracy Using Computerized Adaptive Testing for Mental Health Disorders (CAT-MH). Curr Psychiatry Rep. 2019 Jul 1;21(8):67. doi: 10.1007/s11920-019-1053-9. PMID 31264098
- [Background] Langabeer JR 2nd, Yatsco A, Champagne-Langabeer T. Telehealth sustains patient engagement in OUD treatment during COVID-19. J Subst Abuse Treat. 2021 Mar;122:108215. doi: 10.1016/j.jsat.2020.108215. Epub 2020 Nov 24. PMID 33248863
- [Background] Ryan RM, Deci EL. Self-determination theory and the facilitation of intrinsic motivation, social development, and well-being. Am Psychol. 2000 Jan;55(1):68-78. doi: 10.1037//0003-066x.55.1.68. PMID 11392867

DOCUMENTS (1):
  • Informed Consent Form (2022-12-20): https://cdn.clinicaltrials.gov/large-docs/07/NCT05184907/ICF_001.pdf